CLINICAL TRIAL: NCT04244253
Title: A Randomized, Multi-center, Double-blind, Placebo-controlled, Parallel-group Comparison Trial to Assess Efficacy and Safety of OPC-64005 in Patients With Major Depressive Disorder
Brief Title: A Phase 2 Trial of OPC-64005 for Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 277-102-00027; JapicCTI-205116 (Other: JapicCTI)
Record Dates: First submitted 2020-01-23; First posted 2020-01-28 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- OPC-64005 20 mg (Experimental)
  Interventions: Drug: OPC-64005 20 mg , Once-daily
- OPC-64005 10 mg (Experimental)
  Interventions: Drug: OPC-64005 10 mg , Once-daily
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo, Once-daily

INTERVENTIONS:
Drug: OPC-64005 20 mg , Once-daily — Active, High Dose
  Arms: OPC-64005 20 mg
Drug: OPC-64005 10 mg , Once-daily — Active, Low Dose
  Arms: OPC-64005 10 mg
Drug: Placebo, Once-daily — Placebo
  Arms: Placebo

SUMMARY:
The objective of the trial is to compare the efficacy of OPC-64005 at 20 mg vs placebo and to assess the safety and pharmacokinetics of OPC-64005 at 10 and 20 mg in patients with major depressive disorder (MDD).The primary endpoint is the mean change from baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) total score at Week 6 of the double-blind treatment period in the OPC-64005 20-mg group compared with the placebo group

ELIGIBILITY:
Inclusion Criteria:

* Patients with a DSM-5 classification-based diagnosis of "major depressive disorder, single episode" or "major depressive disorder, recurrent episode" with the current episode persisting for ≥4 weeks to ≤1 year
* Patients with a total score of ≥18 on the 17-item Hamilton Rating Scale for Depression (HAM-D)

Exclusion Criteria:

* Patients with a diagnosis of any of the following diseases according to DSM-5 Neurocognitive disorders, history or complication of schizophrenia spectrum or other psychotic disorder, history or complication of bipolar and related disorders, feeding and eating disorders, obsessive-compulsive disorder, panic disorder, posttraumatic stress disorder, personality disorders, neurodevelopmental disorders, substance-related and addictive disorders (within 180 days prior to informed consent)
* Patients exhibiting mood-incongruent psychotic features in the current major depressive episode
* Patients who, in the opinion of the investigator or subinvestigator, are judged to have treatment-resistant depression, ie, a certain degree of therapeutic effect is not obtained by administration of 2 or more antidepressants having different mechanisms of action at sufficient doses for at least 6 weeks for the current major depressive episode
* Patients receiving augmentation treatment, such as antipsychotics, for the current major depressive episode (excluding the use of sulpiride for depression/depressive state or gastric/duodenal ulcer)

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 273 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Medical Corporation Jisenkai Himorogi Psychiatric Institute, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 273 subjects from 69 trial sites in Japan.
Pre-assignment Details: Adult subjects with Major Depressive Disorder defined by criteria of the Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-5).
Groups:
- OPC-64005 10-mg: One placebo tablet and one OPC-64005 10-mg tablet administered orally once daily for 6 weeks
- OPC-64005 20-mg: One placebo tablet and one OPC-64005 10-mg tablet administered orally once daily for 1 week, followed by two OPC-64005 10-mg tablets for 5 weeks
- Placebo: Two placebo tablets administered orally once daily for 6 weeks
Period: Overall Study
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo
Started | 31 | 121 | 121
Completed | 28 | 116 | 109
Not Completed | 3 | 5 | 12
Not completed — Adverse Event | 2 | 2 | 4
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 6
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set includes all subjects who were administered at least 1 dose of double-blind IMP.
Groups:
- Total: Total of all reporting groups
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo | Total
Number analyzed (Participants) | 31 | 121 | 121 | 273
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 31 | 121 | 121 | 273
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.0) | 39.5 (11.4) | 38.3 (11.1) | 38.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 56 | 58 | 131
  Male | 14 | 65 | 63 | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 31 | 121 | 121 | 273
Region of Enrollment [Number; unit: participants]
  Japan | 31 | 121 | 121 | 273

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score at Week 6 of the Double-blind Treatment Period
Description: The MADRS was a clinician-rated scale which evaluated the level of depression. The MADRS consists of following 10 depressive symptoms on 7 scales of 0 to 6, with higher scores indicating worse condition.
  1. Apparent sadness, 2. Reported sadness, 3. Inner tension, 4. Reduced sleep, 5. Reduced appetite, 6. Concentration difficulties, 7. Lassitude, 8. Inability to feel, 9. Pessimistic thoughts, and 10. Suicidal thoughts
  Summed subscales were combined to compute a total score. Total score ranges form 0 to 60, with higher scores indicating worse condition.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, and 6
Population: The full analysis set (FAS) includes all subjects who were administered at least 1 dose of double-blind IMP and have MADRS total scores at baseline and at least one time point after the start of double-blind treatment. FAS excluded one subject in the placebo group for whom no MADRS total score was obtained after start of double-blind treatment.
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo
Number analyzed (Participants) | 31 | 121 | 120
Units on a scale
  1Week | -1.9 (0.8) | -1.6 (0.4) | -2.1 (0.4)
  2Week: number analyzed (Participants) | 30 | 118 | 119
  2Week | -3.9 (1.0) | -3.4 (0.5) | -3.6 (0.5)
  3Week: number analyzed (Participants) | 29 | 116 | 114
  3Week | -7.1 (1.2) | -5.7 (0.6) | -5.2 (0.6)
  4Week: number analyzed (Participants) | 28 | 116 | 111
  4Week | -9.5 (1.3) | -7.5 (0.7) | -6.3 (0.7)
  5Week: number analyzed (Participants) | 29 | 116 | 109
  5Week | -10.6 (1.4) | -8.9 (0.7) | -8.1 (0.7)
  6Week: number analyzed (Participants) | 28 | 116 | 109
  6Week | -11.2 (1.5) | -10.7 (0.8) | -9.5 (0.8)
Statistical Analysis 1: Comparison: OPC-64005 20-mg vs Placebo; The statistical analysis was performed at Week 6 to compare the OPC-64005 20-mg group and placebo group; Test type: Superiority; p = 0.288, Mixed-model repeated measures; MMRM included treatment, visit, treatment-by-visit interaction, baseline, and baseline-by-visit interaction using an unstructured covariance matrix; Difference of score = -1.1, 95% CI 2-sided [-3.3 to 1.0]

2. Secondary Outcome: MADRS Response Rate
Description: The MADRS response rate is the percentage of subjects with ≥50% reduction from baseline in MADRS total score at Week 6 of the double-blind treatment period.
Time Frame: Baseline, Week 1, 2, 3, 4, 5, and 6
Population: The full analysis set (FAS) included all subjects who were administered at least 1 dose of double-blind IMP and had MADRS total scores at baseline and at least one time point after the start of double-blind treatment.
Measure: Number; unit: percentage of participants
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo
Number analyzed (Participants) | 31 | 121 | 120
percentage of participants
  1Week | 0.0 | 0.8 | 0.8
  2Week | 3.2 | 5.0 | 3.3
  3Week | 12.9 | 9.9 | 6.7
  4Week | 22.6 | 14.9 | 10.0
  5Week | 25.8 | 18.2 | 18.3
  6Week | 32.3 | 29.8 | 24.2
Statistical Analysis 1: Comparison: OPC-64005 20-mg vs Placebo; The statistical analysis was performed at Week 6 to compare the OPC-64005 20-mg group and placebo group; Test type: Other; p = 0.329, χ2 test; The MADRS response rate in the OPC-64005 20-mg group and the placebo group were compared using the χ2 test in the LOCF dataset; Difference in response rate = 5.6, 95% CI 2-sided [-5.6 to 16.8]

3. Secondary Outcome: MADRS Remission Rate
Description: MADRS remission rate is the percentage of subjects with MADRS total score ≤ 10 and ≥ 50% reduction from baseline in MADRS total score at Week 6 of the double-blind treatment period.
Time Frame: Week6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo
Number analyzed (Participants) | 31 | 121 | 120
percentage of participants | 16.1 | 14.9 | 13.3
Statistical Analysis 1: Comparison: OPC-64005 20-mg vs Placebo; The statistical analysis was performed at Week 6 to compare the OPC-64005 20-mg group and placebo group; Test type: Other; p = 0.731, χ2 test; The MADRS remission rate in the OPC-64005 20-mg group and placebo group were compared using the χ2 test in the LOCF dataset; Difference of Proportion = 1.5, 95% CI 2-sided [-7.2 to 10.3]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the date of signed informed consent until 14 (±7) days during the post treatment observation period after the last IMP administration.
Description: An AE is defined as any untoward medical occurrence in a patient or clinical trial subject administered an IMP and which does not necessarily have a causal relationship with this treatment.
Arm/Group | OPC-64005 10-mg | OPC-64005 20-mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/121 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/31 | 2/121 | 1/121
Other Adverse Events (participants affected / at risk) | 7/31 | 19/121 | 19/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-64005 10-mg (N=31) | OPC-64005 20-mg (N=121) | Placebo (N=121)
Appendicitis (Infections and infestations) | 0 | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-64005 10-mg (N=31) | OPC-64005 20-mg (N=121) | Placebo (N=121)
Headache (Nervous system disorders) | 2 | 6 | 3
Insomnia (Psychiatric disorders) | 0 | 8 | 4
Nausea (Gastrointestinal disorders) | 0 | 7 | 9
Nasopharyngitis (Infections and infestations) | 3 | 0 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-03-31): https://cdn.clinicaltrials.gov/large-docs/53/NCT04244253/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT04244253/SAP_001.pdf